CLINICAL TRIAL: NCT04275830
Title: The Effects of Heart Rate Variability Biofeedback Training on Hematopoietic Cell Transplantation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: HonorHealth Research Institute (Other)
Responsible Party: Principal Investigator, Wonsun (Sunny) Kim, Ph.D, Assistant professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00010085; PG12840 (Other Grant/Funding Number: Institute of Social Science Research Center at ASU)
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Hematopoietic Stem Cell Transplantation; Bone Marrow Transplant; Heart Rate Variability; Autonomic Nervous System; Stress; Mood; Psychological Distress; Emotion Regulation; Communication Research; Narrative
Keywords: Digital Storytelling; Narrative; Cancer patients; Bone marrow transplant; Psychosocial health; Heart rate variability biofeedback
MeSH Terms: conditions — Emotional Regulation; Narration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline and HRVB+DS group (Experimental): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture before the random assignment to HRVB+DS arm. This group will receive a standardized HeartMath© Inner balance device and HRV biofeedback training session at the start of the two-week intervention period. They will be asked to attend either a group or one-on-one 30-minute HRVB training session and asked to practice their HRV biofeedback skills at home for 10 minutes each day for a two-week period. Participants will also be asked to watch four digital stories of other HCT patients (2 videos per week) with a weekly email notification and reminder phone call. Each story was made with voice, images, and sound (3-5 minutes each).
  Interventions: Behavioral: Baseline Surveys; Behavioral: Heart rate variability biofeedback
- Baseline and HRVB waitlist +DS control group (Other): In-person baseline surveys using the web-based data collection platform, Research Electronic Data Capture (REDCap) before the random assignment to HRVB waitlist +DS control arm. After the baseline data collection, during two weeks, they will be provided four digital stories of other HCT patients sharing their experiences (challenges, feelings, strategies, coping, each 2-3 minutes long). At the end of the two-week period, participants will be scheduled for a final in-person session including T2 survey and HRV assessment. They will be also provided HRVB training session at T2.
  Interventions: Behavioral: Baseline Surveys; Behavioral: Heart rate variability waitlist and Digital storytelling Control intervention

INTERVENTIONS:
Behavioral: Baseline Surveys — Baseline surveys contained a series of scaled questions, including sociodemographic variables (age, sex, cancer type, and etc), profile of mood states, social well-being, emotional processing and acceptance.
  Other Names: Baseline questionnaire
Behavioral: Heart rate variability biofeedback — Participants randomized to the intervention arm will receive exactly the same four digital stories via REDCap, a standardized HRV sensor and accompanying smart phone app, and a 30-minute HRVB training to use the biofeedback signals to generate a resonant frequency pattern of HRV (coherence) after collecting data at baseline in person. Participants will be given a take-home manual and specifically asked to practice their HRVB skills at home for 5 minutes prior to viewing stories once each week and upload a log of their time practiced to the cloud. The main purpose of adding HRVB practice as a "priming" experience (i.e., to teach participants to practice HRV prior to viewing stories) is to optimize results by focusing patients' and caregivers' skills and experience on HRV as a mechanism of improved emotion regulation, and then combine this achieved coherent pattern with DS intervention.
  Arms: Baseline and HRVB+DS group
Behavioral: Heart rate variability waitlist and Digital storytelling Control intervention — Four Digital Stories Intervention (4 patient stories about hematopoietic cell transplantation (HCT) over the course of 2 weeks (2 videos per week) with a weekly email notification and reminder phone call. Each story was made with voice, images, and sound (3-5 minutes each). The 4 digital stories patients produced contained the following content: (1) a leukemia patient expressed and controlled her depression and anxiety and described how she dealt with the intensive treatment and recovery through a positive attitude and active coping; (2) a mother of 3 children, who was experiencing severe pain due to MS, coped with HCT through family support and positive reframing; (3) a lymphoma patient coped with the HCT procedures by praying during the treatment; and (4) a father of young twins had a HCT twice, and his wife helped him cope with emotional distress through open communication and expressing emotions.Participants will receive a 30-minute HRVB training session at T2.
  Other Names: Narrative-based storytelling
  Arms: Baseline and HRVB waitlist +DS control group

SUMMARY:
Patients undergoing hematopoietic stem cell transplantation (HCT) often continue to experience anxiety, depression, isolation, and other psychosocial distress due to the severe nature of the transplant experience. Storytelling interventions that provide an opportunity for emotional disclosure have shown preliminary efficacy to alleviate psychosocial distress and improve emotion regulation during health challenges. Not only are these changes observed in response to such interventions, but they can also be directly strengthened with HRV biofeedback (HRVB) training, a device-driven breath pacing practice that uses colored light signals to provide feedback to increase vagal tone and improve emotional responses and sleep quality by regulating negative affect and stress. This randomized controlled trial will explore the effects of HRV biofeedback (HRVB) training combined with a digital storytelling intervention and changes in psychosocial distress with a modified waitlist control in a population of Hematopoietic cell transplantation (HCT) patients.

DETAILED DESCRIPTION:
This randomized controlled trial will explore the effects of an HRV biofeedback (HRVB) training session with a modified waitlist control in a population of Hematopoietic cell transplantation (HCT) patients. We will secondarily explore effects of a brief storytelling intervention, with or without the prior HRVB training. Two group of 10 HCT patients over the age of 18 will be recruited and enrolled into the study. The time of participating in this study will be 2-week proposed activities from the time of enrollment to completion. Specific participation will include baseline data collection (about 30 minutes), HRVB training session (30 minutes), watching and discussing stories (15 min for each week= 30 minutes) and one final data collection (about 30 minutes) at the end. For HRVB group, participants will be instructed to practice their HRV biofeedback skills at home for 10 minutes each day for a two-week period (about 140 minutes). Lab visit is required only twice for baseline data collection and final data collection. Other works will be via internet.

ELIGIBILITY:
Patient Inclusion Criteria:

* age 18 or older
* recently underwent Hematopoietic cell transplantation (HCT) (within 3 months after hospital discharge)
* must be able to speak, read, and write in English
* access to a working phone and e-mail account
* have a smart phone

Patient Exclusion Criteria:

* cognitive impairment that prohibits completion of study assessment visual or hearing impairment
* other (e.g., provider non-approval or logistical constraints such as patient moving out of town)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Heart Rate Variability (HRV and coherence scores) at 2 weeks | Baseline (T1), 2 weeks after (T2)
  The Emwave Pro Plus device from HeartMath will be used to collect HRV data and heart rate using a 3-minutes "neutral" protocol (we call "waiting at the bus stop" implying that no particular intent for breath or mindful state is to be evoked) to understand the benefits of DS+ HRVB. In addition, HRV measures will be obtained for the 1-minute paced breathing period to understand the effects of paced breathing on HRV. The following precautions will be provided as instructions to participants prior to data collection: no coffee, tea, or caffeinated drinks such as energizing drinks in the 2 hours before the data collection, and no alcohol consumption during 24 hours prior to the data collection.

SECONDARY OUTCOMES:
Changes from Baseline Profile of Mood States (POMS) short version (Psychological Distress) at 2 weeks | Baseline (T1), 2 weeks after (T2)
  Psychological distress will be measured using the Profile of Mood States (POMS) short version (15 items, 5-point Likert scale; 0=not at all, 4=extremely). The POMS is one of the most frequently used and validated scales in studies of psychosocial interventions for cancer patients. The POMS Total Mood Disturbance (TMD) score has been shown to be most sensitive to interventions designed to facilitate emotional expression. The POMS consists of the TMD dimensions (tension-anxiety; depression-dejection; anger-hostility; and confusion-bewilderment) (Cronbach's a = .93) to be used in the current study as the primary outcome measure; and two others (fatigue-inertia; vigor-activity) will be documented. Total of Mood Disturbance= (anxious+depression+anger+fatigue)- vigor (Range from 12 to 48). The higher values represent a worse emotional well-being.

OTHER OUTCOMES:
Changes from Baseline Depression at 2 weeks | Baseline (T1), 2 weeks after (T2)
  Depression will be measured using the Center for Epidemiological Studies Depression Scale Revised (CESD-R-10) scale (10 items, 4-point Likert scale (0 = rarely or none of the time, 3= all of the times, Cronbach's a = .86). The higher values represent a worse depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Kim, PhD, Principal Investigator — Arizona State University
Locations (1):
- HonorHealth, Scottsdale, Arizona, United States